CLINICAL TRIAL: NCT01183897
Title: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Primary Refractory Neuroblastoma in Bone Marrow: A Phase II Study
Brief Title: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Primary Refractory Neuroblastoma in Bone Marrow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-161
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2018-09

CONDITIONS: Neuroblastoma
Keywords: GM-CSF; MAB 3F8; RETINOIC ACID (CIS-9 & 13); 09-161
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic (Experimental): This phase II study of the anti-GD2 murine IgG3 monoclonal antibody 3F8 combined with granulocyte-macrophage colony stimulating factor (GM-CSF) will assess response in of primary refractory neuroblastoma in bone marrow (i.e., incomplete response to standard treatment).
  Interventions: Biological: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic

INTERVENTIONS:
Biological: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic — This phase II, open-label, single arm trial assesses the anti-NB activity of high-dose 3F8 (80 mg/m2/day), which is used in cycles 1-2, with return to standard 3F8 dosage (20 mg/m2/day) in subsequent cycles.Clinical results will be compared to those in the predecessor trials which used only the standard 3F8 dosage. Starting with A(6), patients no longer receive high-dose 3F8 but receive only standard dose 3F8 (20mg/m2/day) for all cycles The patients have primary refractory BM disease. Protocol treatment is through 24 months.
  Real-time quantitative RT-PCR63-65 will be used to assess MRD in BM. 13-cis-retinoic acid is started no later than after cycle 4 (i.e., after response is scored), but sooner if CR is achieved after cycles 1, 2, or 3, or if early HAMA develops.

SUMMARY:
The purpose of this study is to see find out what effects, good and/or bad, the combination of 3F8 and GM-CSF has on the patient and the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by a) histopathology (confirmed by the MSKCC Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels.
* High-risk NB as defined by risk-related treatment guidelines1 and the International NB Staging System,89 i.e., stage 4 with (any age) or without (> or = to 18 months of age) MYCN amplification or MYCN-amplified stage 4S.
* Patients have primary refractory disease limited to BM, i.e., high-risk NB (defined above) resistant to standard therapy, as evidenced by incomplete response in BM, but no measurable MIBG-avid soft tissue tumor assessable for response and no progressive disease.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Creatinine > 3.0 mg/dL
* ALT, AST and Alkaline Phosphatase > 5.0 times the upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with grade 3 or higher toxicities (using the CTCAE v 4.0) related to cardiac, neurological, pulmonary or gastrointestinal function as determined by physical exam. Patients must have normal blood pressure for age.
* Progressive disease
* History of allergy to mouse proteins.
* Active life-threatening infection.
* Human anti-mouse antibody (HAMA) titer >1000 Elisa units/ml.
* Inability to comply with protocol requirements.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Modak S, Basu EM, Roberts SS, Kramer K, Cheung NK. Posterior reversible encephalopathy syndrome in neuroblastoma patients receiving anti-GD2 3F8 monoclonal antibody. Cancer. 2013 Aug 1;119(15):2789-95. doi: 10.1002/cncr.28137. Epub 2013 Apr 30. PMID 23633099
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 28
  Greece | 1
  Israel | 2

OUTCOME MEASURES:

1. Primary Outcome: Assess the Activity of High-dose 3F8/GM-CSF
Description: against persistent neuroblastoma in bone marrow of patients who have no other evidence of disease by standard studies.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic
Number analyzed (Participants) | 0

2. Secondary Outcome: Apply Real-time Quantitative RT-PCR
Description: to test the hypothesis that the minimal residual disease content of bone marrow after the first treatments with 3F8/GMCSF has significant prognostic impact on progression-free survival.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic
Number analyzed (Participants) | 0

3. Secondary Outcome: Monitor Safety of the High-dose Antibody Treatment
Description: to assure no side-effects or noxious sequelae develop or emerge that were not seen in the prior phase I study.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Data were not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT01183897/Prot_SAP_000.pdf